CLINICAL TRIAL: NCT01843309
Title: Use of Spironolactone for the Prevention of Electrolyte Abnormalities in Patients Treated With Amphotericin B
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not possible to complete the sample within the estimated time by the use of new antifungals
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Bertha Manuela Córdova Sánchez, Fellow, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AMPHYRO-628
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Patients With Fungic Infections
MeSH Terms: interventions — Canrenoic Acid; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Spironolactone 200mg (Experimental): Spironolactone 100 mg twice a day orally
  Interventions: Drug: Spironolactone 200mg
- Placebo (Placebo Comparator): Placebo twice a day orally
  Interventions: Drug: Placebo
- Spironolactone 100mg (Experimental): Spironolactone 100mg once a day
  Interventions: Drug: Spironolactone 100mg

INTERVENTIONS:
Drug: Spironolactone 100mg
  Arms: Spironolactone 100mg
Drug: Spironolactone 200mg
  Arms: Spironolactone 200mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Purpose Invasive fungal infections cause significant morbidity and mortality in immunocompromised patients.

Amphotericin B deoxycholate (AmB) is a polyene antifungal agent. The broad spectrum of activity contributed to it being considered the gold standard of antifungal therapy despite being associated with high incidences of infusion related adverse events.

AmB exerts their antifungal effect binding to ergosterol; a sterol similar to cholesterol found in fungal cell membranes. However AmB also binds to cholesterol molecules in mammalian cell membranes forming intramembranous pores and vacuoles in the distal convoluted tubule of the kidney producing its nephrotoxic effects.

Nephrotoxicity is the major adverse effect of AmB, often limiting administrations of full dosage; it's manifested as acute kidney injury, impaired renal concentrating ability, augmented urinary potassium secretion through tubular Na+/K+ ATPase, type-1 renal tubular acidosis, which increases the elimination of potassium, and magnesium wasting. Furthermore potassium depletion potentiates the tubular toxicity of AmB.

The management of potassium wasting may be difficult, even high intravenous doses of potassium chloride may not be fully effective in correcting the hypokalemia. It has been probed the use of potassium-sparing diuretics to limit electrolyte wasting in patients treated with AmB.

In 1988 Smith et al, demonstrated that amiloride was well tolerated and provided effective control of plasma potassium in patients treated with AmB. This finding was confirmed in 2001 by Bearden et al. However in our country the only available commercial presentation of amiloride also contains hydrochlorothiazide, limiting its use in such patients.

Spironolactone acts on the distal renal tubule by competitive inhibition of aldosterone, thereby blocking the exchange between sodium and both potassium and hydrogen in the distal tubules and collecting ducts. These agents produce a sodium diuresis which results in potassium retention. There is only one clinical trial by Ural et al, using spironolactone to prevent hypokalemia in twenty-six neutropenic patients on AmB treatment; they demonstrated that those patients receiving concomitant AmB and spironolactone (100mg bid) had significantly higher plasma potassium levels than those receiving AmB alone (P=0.0027) and required significantly less potassium supplementation to maintain their plasma potassium within the normal range (P=0.022).

Renal vasoconstriction appears to play a major role in AmB induced reduction in GFR; recurrent ischemia may lead to structural and tubular damage and permanent nephrotoxic effects.

Aldosterone modulates the tone of the renal vasculature. Bobadilla et al have shown in animal models of cytotoxic damage using cyclosporine; that a mineralocorticoid receptor blockade with spironolactone reduces the structural renal damage, and also prevents renal dysfunction due to afferent and efferent vasoconstrictions. This group has also shown that prophylactic treatment with spironolactone completely prevents renal dysfunction and histological signs of tubular injury from ischemia-reperfusion injuries. And also has demonstrated the ability of spironolactone in animal models to protect the kidney after establishing an ischemic insult, when spironolactone was administrated immediately or 3h after the renal ischemic insult had occurred, reducing levels of sensitive biomarkers such as Kim-1 and Hsp70.

The investigators' hypothesis is that administration of spironolactone in patients treated with AmB will help to maintain significantly higher plasma potassium levels and will help to reduce potassium and magnesium supplementation. Moreover spironolactone will help to reduce the urinary excretion of potassium.

The investigators propose a randomized, double blind, placebo controlled trial approved by the local ethical committee, to compare the efficacy and security of spironolactone to reduce electrolytic derangements in three groups: AmB and placebo, AmB and spironolactone 100mg once a day, AmB and spironolactone 100mg twice a day. The investigators will include 12 patients per group. Researchers will collect daily plasma creatinine, sodium, potassium, BUN and urinary potassium, as well as the values of potassium and magnesium supplements administered orally or parenterally. The researchers will also collect by 7 days urinary levels of NGAL, KIM-1 and Hsp-70 as tubular injury markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indications for AmB treatment

Exclusion Criteria:

* Patients with acute kidney injury
* Hyperkalemia ≥5.2
* Hypersensibility to spironolactone
* HIV infection
* Pregnant women
* Solid organ transplant
* Hemodynamic instability
* CKDEPI ≤30ml/min/1.73m3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of hypokalemia ≤3.5mEq/L | Up to the 5th day
  Researchers will collect daily plasma potassium
Average potassium supplementation | Within the first to 15 days
  Researchers will collect the values of potassium supplements administered orally or parenterally.
Incidence of hyperkalemia | Up to the 5 day
  Researchers will collect daily plasma potassium levels.

SECONDARY OUTCOMES:
Acute kidney injury | Within the first 15 days
  Researchers will collect daily plasma creatinine and urinary output. We will define acute kidney injury by creatinine elevation ≥0.3mg/dL above de baseline or reduction in urinary output according to AKIN criteria.
Incidence of renal tubular damage | Up to the 7th day
  Researchers will also collect by 7 days urinary levels of NGAL, KIM-1 and Hsp-70 as tubular injury markers.
Incidence of hypomagnesemia | Up to the 15 day
  Researchers will collect daily plasma magnesium

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, México, State of Mexico, Mexico